CLINICAL TRIAL: NCT01253447
Title: A Phase 2 Study of the AKT Kinase Inhibitor MK-2206 in Patients With Relapsed Refractory Acute Myelogenous Leukemia
Brief Title: AKT Inhibitor MK-2206 in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2010-02186; NCI-2010-02186 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2010-0243 (Other: M D Anderson Cancer Center); 8731 (Other: CTEP); N01CM00039 (NIH); NCT01654978 (obsolete NCT alias)
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — MK 2206

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Akt inhibitor MK2206) (Experimental): Akt inhibitor MK2206 200 mg orally once a week for each 28 day treatment cycle
  Interventions: Drug: Akt inhibitor MK2206; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Akt inhibitor MK2206 — 200 mg orally (PO) once weekly. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: MK2206
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well AKT inhibitor MK-2206 works in treating patients with relapsed or refractory acute myeloid leukemia (AML). AKT inhibitor MK-2206 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the proportion of patients achieving Morphologic Complete Response (CR), Morphologic CR with incomplete count recovery (CRp) or Partial Response (PR) as best response within 3 cycles of therapy with MK-2206.

SECONDARY OBJECTIVES:

I. Describe the disease-free survival of patients that achieve CR/CRp.

II. Determine the toxicity profile of single-agent MK-2206 in this patient population.

III. To determine the biologic effects of MK-2206 on leukemia cells.

OUTLINE:

Patients receive AKT inhibitor MK-2206 orally (PO) once weekly. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed AML other than acute promyelocytic leukemia (2008 World Health Organization (WHO) classification)
* Patients must have persistent or relapsing disease requiring 2nd salvage therapy (e.g. treatment for second or higher relapse or for primary refractory disease after failure of two prior treatment regimens); duration of prior complete remission < 12 months if not refractory disease; patients with prior autologous and allogeneic hematopoietic stem cell transplantation are eligible if patients are off immunosuppression for >1 month and have no evidence of active graft versus host disease (GVHD) except grade 1 skin GVHD
* Patients age >= 60 years with less than two prior treatment regimens not candidates for or have refused standard chemotherapy, excluding subjects with acute promyelocytic leukemia (APL) or with favorable cytogenetic abnormalities [inv16, t(8;21)]
* Patient at the time of enrollment should not be a candidate for allogeneic stem cell transplantation
* The Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Serum creatinine or calculated creatinine clearance =< 1.5 * upper limit of normal (ULN) OR >= 60 mL/min for patients with creatinine levels > 1.5 * institutional ULN
* Serum total bilirubin =< 2 * ULN OR direct bilirubin =< ULN for patients with total bilirubin levels > 2 * ULN, unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis
* asparate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT /SGPT) =< 2.5 * ULN or =< 5 * ULN unless considered to be secondary to leukemic involvement
* Fasting serum glucose =< 150 mg/dl
* HBA1c =< 9%
* Female patient of childbearing potential must have a negative serum or urine pregnancy test beta- Human chorionic gonadotropin (hCG) within 72 hours prior to receiving the first dose of study medication; the effects of MK-2206 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason women of childbearing potential and men must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treatment physician immediately
* Patient, or the patient"s legal representative, has voluntarily agreed to participate by giving written informed consent
* Patient is able to swallow tablets and has no surgical or anatomical condition that will preclude the patient from swallowing and absorbing oral medications on an ongoing basis

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery
* Active uncontrolled infection
* Systemic chemotherapy (with the exception of hydroxyurea) within 14 days (or within 5 half-lives for an investigational agent) prior to first dose of study drug, unless there is evidence of rapidly progressive disease; persistent chronic clinically significant toxicities from prior chemotherapy must not be > grade 1
* Patients with central nervous system (CNS) involvement
* Patient has known hypersensitivity to the components of study drug or its analogs
* Uncontrolled congestive heart failure, unstable angina pectoris
* Uncontrolled cardiac arrhythmia
* History or current evidence of a myocardial infarction during the last 6 months
* corrected Q-T interval (QTc) prolongation > 450 msec (Bazett's Formula)
* Congenitally long QT syndrome, has received any marketed or experimental compound in the last 4 weeks or 5 half lives (whichever is shorter) prior to entering the study with possible or known effects of QT prolongation
* Patient with symptomatic bradycardia, or a history of clinically significant bradyarrhythmias such as sick sinus syndrome, 2nd degree AV block (Mobitz Type 2)
* Patient with uncontrolled hypertension (i.e., i.e., sustained systolic blood pressure >= 160 or diastolic >= 90); patients who are controlled on antihypertensive medication will be allowed to enter the study
* Patient with poorly controlled diabetes defined as HBA1C > 9%
* Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study
* Patient is known to be Human Immunodeficiency Virus (HIV)-positive with history of AIDS defining conditions; or CD4 cells prior to leukemia onset =< 400 cells/mm^3; or patients receiving antiretroviral therapy that affects CYP3A4 such as protease inhibitors, efavirenz, nevirapine, or zidovudine
* Patient has active Hepatitis B or C or active Hepatitis A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Konopleva, MD, PHD, Principal Investigator — UT MD Anderson Cancer Center
Locations (2):
- United States (2):
  - UT MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Konopleva MY, Walter RB, Faderl SH, Jabbour EJ, Zeng Z, Borthakur G, Huang X, Kadia TM, Ruvolo PP, Feliu JB, Lu H, Debose L, Burger JA, Andreeff M, Liu W, Baggerly KA, Kornblau SM, Doyle LA, Estey EH, Kantarjian HM. Preclinical and early clinical evaluation of the oral AKT inhibitor, MK-2206, for the treatment of acute myelogenous leukemia. Clin Cancer Res. 2014 Apr 15;20(8):2226-35. doi: 10.1158/1078-0432.CCR-13-1978. Epub 2014 Feb 28. PMID 24583795
- See also: UT MD Anderson Cancer Center Official Website — http://www.mdanderson.org
- See also: Fred Hutchinson Cancer Research Center Official Website — http://www.fhcrc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 27, 2010 to October 30, 2012. All recruitment done in medical clinics, either UT MD Anderson Cancer Center or Fred Hutchinson Cancer Research Center.
Period: Overall Study
Arm/Group | Treatment (Akt Inhibitor MK2206)
Started | 19
Completed | 17
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 72 [31 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response of CR, CRp, or PR
Description: Responses defined by International Working Group (IWG) 2003 Response Criteria: Morphologic Complete Response (CR): Peripheral blood counts: No circulating blasts, Neutrophil count >/= 1.0 x10^9/L, Platelet count >/= 100 x10^9/L; Bone marrow aspirate and biopsy: </= 5% blasts, No detectable Auer rods, No extramedullary leukemia. Partial Response (PR): No circulating blasts, Neutrophil count >/=1.0 x10^9/L, Platelet count >/= 100 x10^9/L, >/= 50 % reduction in bone marrow blast to 6% to 25%, or blasts </= 5% if Auer rods are present. Morphologic CR with incomplete count recovery (CRp): All criteria for CR except for residual neutropenia (<1x10^9/L) or thrombocytopenia (<100 x10^9/L).
Time Frame: 12 weeks of treatment
Population: No participant was not evaluable for response.
Measure: Number; unit: participants
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 18
participants
  CR | 0
  CRp | 1
  PR | 0

2. Primary Outcome: Number of Participants With Treatment-related Non-hematological Toxicity
Description: Toxicity assessed using the NIH-NCI Common Terminology Criteria for Adverse Events, version 4.0 (CTCAEv4.0)
Time Frame: Up to 30 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 18
Participants
  Neutropenic Fever | 2
  Documented infection | 6
  Pneumonia | 2
  Fever of Unknown Origin | 2
  QTc Prolongation | 4
  Maculopapular Rash | 10
  Hyperglycemia | 12
  Posterior reversible encephalopathy (PRES Syndrome | 1

3. Secondary Outcome: Maximum Percentage Change in Apoptosis
Description: Peripheral blood Acute Myeloid Leukemia (AML) cells (total 2 x 10^6) used to determine induction of apoptosis in AML stem cells by 4-color flow cytometry assay (CD34/CD38/CD123/annexin). Two-sample t-test conducted to compare changes between the responders and non-responders. Responders are participants who obtain a CR, CRp, or PR, with or without cytogenetic response.
Time Frame: Baseline to 12 courses
Population: The Assay did not work so no comparison can be made.
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants followed for up to a total of 12 cycles (up to 36 weeks), with serious adverse events captured from consent until 30 days after last dose of drug. Overall adverse events were collected from January 26, 2011 to October 22, 2012.
Arm/Group | Treatment (Akt Inhibitor MK2206)
Serious Adverse Events (participants affected / at risk) | 12/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=19)
Anorectal infection (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Febrile neutropenia (Infections and infestations) | 5 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections (Infections and infestations) | 2 (2) — Lung, Sepsis
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Symptoms skin lesions
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Pain in extremity (Investigations) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Bilateral carck in lungs (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Mucor fungal infection (Skin and subcutaneous tissue disorders) | 1 (1)
Soft Tissue Infection (cellulitis) (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=19)
Anorexia (Gastrointestinal disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2)
Chills (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine increased (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (11)
Dizziness (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Edema limbs (Blood and lymphatic system disorders) | 3 (3)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1)
Hidradenitis (Endocrine disorders) | 1 (1)
Epistaxis (General disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 8 (8)
Fever (Investigations) | 3 (3)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1 (1)
Poor Appetitue, Gastrointestinal (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (26)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Throat Yeast infection (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Pancytopenia (Investigations) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 2 (5)
Periorbital edema (Eye disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (6)
acute renal insufficiency, elevated creatinine (Renal and urinary disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (3)
Leukemia Cutis (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less